CLINICAL TRIAL: NCT03986216
Title: Development of a Portable Synergy Resistant EMG-driven FES Device for Intuitive Control of Grasp and Release During Functional Arm Activities Following Stroke
Brief Title: Development of a FES Device for Hand Use During Arm Activities Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jun Yao, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00072008
Record Dates: First submitted 2019-05-01; First posted 2019-06-14 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Hand Function
Keywords: Stroke rehabilitation; Hand opening; Functional electrical stimulation; Home-based intervention; Task-specific practice; Device-assisted practice
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a small clinical trial to determine the feasibility of the product for the purpose of home-based arm/hand practice. We will recruit 2-4 stroke participants to participate the small clinical trial (i.e., the home based practice).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Home based group (Experimental): This group will involve 2-4 randomly selected participants who have already completed the lab based sessions. They will use the developed reliable and intuitive control of the paretic hand device (ReIn-Hand device) to assist them to practice 'reach-grasp-retrieve-release' movements at home, 1 hours per day (20 trials), 7 days per week for 12 weeks.
  Interventions: Device: ReIn-Hand device assisted home-based practice

INTERVENTIONS:
Device: ReIn-Hand device assisted home-based practice — Practice reach-grasp-retrieve-release at home with the aid of ReIn-hand device

SUMMARY:
The goal of the study is to develop an individualized, synergy resistant, portable electromyographic (EMG)-driven functional electrical stimulation (FES) device that allows for Reliable and Intuitive control of hand (ReIn-Hand) opening while using the paretic arm during lifting and reaching. Furthermore, to enable sufficient practice intensity both in the clinic and at home, the investigators propose to develop the ReIn-Hand device with easy-to-use utilities by developing a user-customized forearm/hand orthosis with embedded EMG recording and stimulation electrode. To test the device feasibility, a small clinical trial will be conducted. Information related to the clinical trial will be provided below.

DETAILED DESCRIPTION:
Individuals with moderate to severe stroke will be recruited for both lab-based testing and home-based practice:

1. Pre-training clinical evaluation (lab-based). In this session, a research physical therapist will evaluate the participant's arm function and impairment level using standardized clinical assessments to ensure eligibility for participating in this study. Once confirmed, a set of standardized clinical assessments will be conducted by the research physical therapist as the baseline assessments of the participant's hand/arm function. This visit is expected to last approximately 3 hours.
2. Pre-training device setup (lab-based). The participant will be randomly assigned to one of the recruited physical therapists (PTs) or senior student physical therapists (SPTs) who has been recruited and consented to participate in this study. The assigned PT will determine 1) the electrode positions for recording the participant's muscle activities during the performance of different arm/hand functions, and 2) the stimulation electrode positions and stimulation intensities for achieving the best hand opening with the forearm at the individual's mid-range of available supination/pronation. Then, the corresponding electrode positions will be marked, and the forearm/hand with these markers will be scanned. This visit is expected to last approximately 3 hours. The scanned results will be used offline to develop a forearm-hand orthosis (FHO) that fits the participant's forearm and hand. During this visit, the investigators will measure the time for the PT/SPT to set up 1) recording electrodes, 2) detecting rules, 3) stimulation electrodes and configuration, and 4) the time for scanning.
3. Pre-training device-use learning sessions (2 visits, lab-based). After the FHO is ready, the participant will be called to participate in the 1st and 2nd lab-based training sessions for the use of ReIn-hand device. During these 2 visits, the assigned PT/SPT (1st test) or the research PT (2nd test) will train the participant to use the FHO and the ReIn-Hand software on a mobile device, until the participant demonstrates the ability in using the device independently twice in a row. During these 2 visits, the investigators will measure the time for the participant to 1) learn the use of the ReIn-Hand device (from the start of the session to the time that the participant is able to demonstrate ability to independently use the device twice in a row), 2) attach the FHO, 3) use the software for 1 trial (including connecting all the cables following the instructions, start the software and finish 1 trial), and 4) clean up. At the end of the 1st (for PTs) or the 2nd (for individuals with stroke) learning sessions, a 5min user survey will be conducted to report the level of ease-of-use of the ReIn-Hand device. During the 2nd learning session, the participant will also be re-tested on part of the clinical assessments, however, this time with the assistance of the ReIn-Hand device. Each of these 2 visits is expected to last about 3 hours.
4. Pre-training 2nd baseline clinical measures (lab-based). Within one week prior to starting the Home-based practice, a research PT will conduct the 2nd baseline clinical measures, which will repeat the 1st baseline clinical measures with an additional quantitative measure of maximal hand opening area and closing force (QMHOC). For QMHOC, pressure sensors (Pressure Profile Systems, Inc., Los Angeles, CA 90045) in conjunction with portable Moire Phase Tracking cameras (Metria Innovation, Inc., Wauwatosa, WI) will be used. The whole QMHOC will take about 10 minutes, and the whole 2nd baseline clinical measure session will take about 2 hours.
5. Pre-training EEG measures (lab-based). Within one week prior to starting the Home-based practice and within one week following completion of the 12-week Home-based practice, the participant will take part in an EEG experiment. During this session, a 9x9 mm marker will be placed on the tip of each finger, with another on the back of the hand as reference, which will allow for the measure of the position and angle of the fingers/hand by 2 portable Moire Phase Tracking cameras (180 Hz; Metria Innovation Inc. Milwaukee, WI). In addition, surface EEG electrodes will be mounted on a stretchable fabric cap based on the 10/20 system. A Polaris Krios handheld scanner and reflective markers (NDI, Ontario, Canada) will be used to record the EEG electrode positions compared to the coordinate system defined by the nasion, inion, and pre-auricular notches. Eye movement detection electrodes will also be placed on the supra- and infra-orbital margins for detection of vertical eye movement. EMG will be recorded from the extensor carpi radialis, flexor carpi radialis, and deltoid of the arm.

   Once prepared, the participant will be seated in an experimental chair with: 1) adjustable straps across the shoulders and waist to maintain proper posture, 2) paretic forearm attached to an orthosis that is linked to the Arm Coordination Training 3D robot(ACT-3D), a robot that will provide required arm support, 3) hand around a cylinder with a custom pressure sensor mat (Pressure Profile System Inc., CA). The participant will be instructed to perform 1 of 2 movements: 1) hand opening while resting on a haptic table, or 2) hand opening while lifting against 50% of their maximum shoulder abduction force. The investigator will measure scalp recordings and EMG recordings using a 160-channel EEG/EMG system using active electrodes (Biosemi, Inc., Active II, Amsterdam, The Netherlands), hand opening area or finger flexion force.
6. Home-based practice. After above 5 lab-based visits, participants will take the ReIn-Hand device, including the FHO, the mobile device with ReIn-Hand software, and the electronic stimulator (EMPI 300PV, Minnesota, USA, a FDA approved clinical device) back home. At home, participants will perform 20 trials of pre-set tasks, like reaching and grasping, per session (1 hour), 1 session per day, 7 days per week for 12 weeks. During these 12 weeks, the participant will visit the lab once per week to make necessary device changes, and perform part of the clinical assessments and QMHOC measure without the ReIn-hand.
7. Post-training tests (lab-based). The sessions #4 mentioned above will be repeated at one week and 3-month after the 12-week home-based practice. The session #5 will be repeated at one week after the 12-week home-based practice. All the post-training tests will be preformed without ReIn-hand device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-80
* Paresis confined to one side, with substantial motor impairment of the upper limb and some residual voluntary movement (Upper Extremity Fugl-Meyer Assessment (UEFMA) in the range of 10-40/66, Chedoke McMaster Stroke Assessment Hand (CMSA_H) stage of the hand section <=4)
* Normal Cognitive ability (MOCA score >=24)
* Capacity to provide informed consent
* Ability to elevate their limb against gravity up to at least 75 degrees of shoulder flexion and then to generate some active elbow extension
* Ability to open hand with a thumb-to-index finger distance ≥4 cm, with the assistance of the ReIn-Hand device with the help of a physical therapist
* Discharged from all forms of physical rehabilitation
* Intact skin on the hemiparetic arm

Exclusion Criteria:

* Motor or sensory impairment in the non-affected limb
* Any brainstem and/or cerebellar lesion
* Severe concurrent medical problems (e.g. cardiorespiratory impairment, uncontrolled hypertension, inflammatory joint disease)
* History of neurologic disorder other than stroke (Parkinson's Disease, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Traumatic Brain Injury, peripheral neuropathy)
* Any acute or chronic painful condition in the upper extremities or spine, indicated by a score ≥5 on a 10-point visual analog scale
* Using cardiac pacemaker
* Seizure
* Severe upper extremity sensory impairment indicated by absent sharp-blunt discrimination on the tactile sensation subscale of the Revised Nottingham Sensory Assessment( the score >=1 on anterior and posterior forearm)
* Chemo denervation: botulinum toxin injection to any portion of the paretic UE within the last 6 months, or phenol/alcohol injections <12 months before participation
* Unable to passively attain 90 degrees of shoulder flexion and abduction, measured using a goniometer based on adapted methods
* Flexion contractures larger than 30 degrees in the elbow, wrist, metacarpophalangeal joints (MCP) and interphalangeal joints (IP)
* Pregnant or planning to become pregnant
* Upper extremity musculoskeletal impairment limiting function prior to stroke.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yao, PhD, Principal Investigator — Department of Physical Therapy and Human Movement Sciences, Northwestern University
Locations (1):
- Northwestern University, Dept. of PTHMS, Chicago, Illinois, United States

REFERENCES:
- [Derived] Carmona C, Sullivan JE, Arceo R, Drogos J, Besser S, Gutierrez S, Jeteric Z, Wyman J, Yao J. Development and Preliminary Validity Study of a Modified Version of the Upper Extremity Fugl-Meyer Assessment for Use in Telerehabilitation. J Neurol Phys Ther. 2023 Oct 1;47(4):208-216. doi: 10.1097/NPT.0000000000000447. Epub 2023 Jun 14. PMID 37314323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DEV14 on 5/17/2019 DEV43 on 12/17/2019 DEV201 on 7/22/2020
Pre-assignment Details: No significant events.
Groups:
- Home Based Group: This group will involve 2-4 randomly selected participants who have already completed the lab based sessions. They will use the developed ReIn-Hand device to assist them to practice 'reach-grasp-retrieve-release' movements at home, 1 hours per day (20 trials), 7 days per week for 12 weeks.
  ReIn-Hand device assisted home-based practice: Practice reach-grasp-retrieve-release at home with the aid of ReIn-hand device
Period: Overall Study
Arm/Group | Home Based Group
Started | 3 (DEV14 1st baseline on 7/16/2019)
Completed | 3 (3-m followup on DEV201 on 3/18/2021)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Three chronic (>1y) post-stroke subjects who suffers single side stroke with moderate to severe impairment (FMA baseline ranging 27-35), CheDock 3-4) participated the home-based intervention.
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.33 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/non-hispanic | 2
  African American/non-hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Box and Blocks [Mean (Full Range); unit: blocks] — The individual is instructed to move as many blocks as possible, one at a time, from one compartment to another for a period of 60 seconds. The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other. Patients hand must cross over the partition in order for a block to be counted, and blocks that drop or bounce out of the second compartment onto the floor are still rewarded with a point. Multiple blocks carried over at the same time count as a single block. The reported results have decimals since we take the mean of 2 baseline assessments.
  blocks | 13.74 [6 to 19.5]
Action Research Arm Test (ARAT) [Mean (Full Range); unit: scores on a scale] — The Action Research Arm Test (ARAT) is a measure consisting of 19 items. There are 4 subscales (grasp, grip, pinch, and gross arm movement). The possible scale range for each item is 0 to 3:
  0 - can perform no part of the test
  1. - performs test partially
  2. - completes test, but takes abnormally long or has great difficulty
  3. - performs test normally
  Subscales are summed to get a participant's total score. The minimum total score is 0, and the maximum total score is 57. Higher values indicate better performance. Reported score has decimals as it is the average of 2 baseline assessments.
  scores on a scale | 29.6 [20.5 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Box and Blocks Test (BBT) Score Across the 12 Weeks of the Intervention, Immediately After Conclusion of Intervention, and 3 Months Post-intervention
Description: Individuals are seated at a table, facing a rectangular box that is divided into two square compartments of equal dimensions by means of a partition. One hundred and fifty small wooden cubes or blocks are placed in one compartments or the other. The individual is instructed to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds. The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one minute trial period. Patients hand must cross over the partition in order for a point to be given, and blocks that drop or bounce out of the second compartment onto the floor are still rewarded with a point. Multiple blocks carried over at the same time count as a single block. The reported results have decimals since we take the mean of 2 baseline assessments.
Time Frame: Assessed at baseline, weekly during intervention, post-intervention (within 1 week after conclusion of intervention), and 3 month follow up (assessed for up to 6 months total); baseline, post-intervention and 3 month follow up (6 months) data reported.
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side.
Measure: Mean (Full Range); unit: blocks
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
blocks
  baseline | 13.74 [6 to 19.5]
  post-intervention | 21 [14 to 27]
  3m follow-up | 19.67 [17 to 24]

2. Secondary Outcome: Upper Extremity Fugl-Meyer Assessment Motor (FMA) Score
Description: The Fugl-Meyer Assessment of Motor Recovery after stroke evaluates and measures recovery in post-stroke hemiplegic patients. It is used in both the clinical and research settings, and is one of the most widely used quantitative measures of motor impairment. Areas of assessment include activities of daily living, functional mobility, and pain. Different movements are judged on the individuals ability to perform with full capacity, limited capacity, or total inability to complete the movement. Scores range from 0-66, with 0 and 66 representing no and normal residual upper extremity motor function, respectively. Higher scores indicate a better outcome.
Time Frame: Assessed at and data presented and reported for baseline, post-intervention (within 1 week after last intervention), and at a 3 month follow up (assessed for up to 6 months total).
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Upper Extremity Fugl-Meyer Assessment Motor (FMA) Score for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  baseline | 31.83 [29 to 35]
  post-intervention: number analyzed (Participants) | 2
  post-intervention | 38 [38 to 38]
  3m follow-up | 36.33 [30 to 40]

3. Secondary Outcome: Quantitative Measure of Hand Opening Area and Closing Force
Description: Individual will be instructed to rest paretic hand on a cylinder that is covered with an array of pressure sensors (Pressure Profile Systems, Inc., Los Angeles, California 90045). Furthermore, 5 markers (9x9 mm) with unique optical features will be placed on the tip of the thumb and the 4 fingers. Individual will then be instructed to perform following task in their comfortable pace: 1) resting, 2) maximally open the paretic hand, and 3) maximally close the paretic hand against the cylinder. Position (with an accuracy of 1mm) and angular (with an accuracy at 0.02 degree) information of fingertips will be captured by 2 registered portable Moire Phase Tracking cameras (Metria Innovation, Inc., Wauwatosa, WI); and the flexion force under the 4 fingers and thumb will be measured by the pressure sensors. This will allow for tracking of the hand pentagon area and closing force during intervention.
Time Frame: This will be measured pre-intervention (within 1 week prior to intervention), 1 time per week during intervention, immediately after conclusion of intervention (within 1 week), and at a 3 month follow up
Population: Data could not be collected safely for 2 subjects due to restrictions from the Coronavirus Disease of 2019 (COVID-19) pandemic. The data collected for the first subject was of poor quality and could not be analyzed.
Arm/Group | Home Based Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Sensory Assessment (Stereognosis)
Description: Stereognosis refers to the ability to identify or perceive the material quality of objects through touch alone, in the absence of visual or auditory stimuli. The individual will be asked to use their paretic hand to identify a number of everyday items through touch alone. Scores range from 0-24, with 24 indicating full stereognosis function and 0 representing complete absence of stereognosis. Decimals are included in the lower and upper limits of the Full Range in the "baseline" row as these resulted from the averaging of two baseline scores.
Time Frame: as for outcome 2
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Sensory Assessment (Stereognosis) Score for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  Baseline | 13.83 [2.5 to 21.5]
  Post-intervention: number analyzed (Participants) | 2
  Post-intervention | 12.5 [3 to 22]
  3m follow-up | 15.33 [3 to 22]

5. Secondary Outcome: Cutaneous Sensory Touch Threshold Using Semmes-Weinstein Monofilaments
Description: The monofilament test is a threshold assay used to determine the minimum force that can be felt by a subject. This test is also known as light touch/protective touch/deep pressure testing in the hands. There are 6 monofilament sizes used to test, with each having a corresponding target force in grams. They are as follows, with the target force in grams in parentheses:
  2.83 (0.07) - Normal 3.61 (0.4) - Diminished Light Touch 4.31 (2) - Diminished Protective Sensation 4.56 (4) - Loss of Protective Sensation 5.07 (10) - Loss of Protective Sensation 6.65 (300) - Deep Pressure Sensation only
  6 parts of the hand were tested. These 6 values were then averaged. The minimum score for the test is 2.83 and the maximum score is 6.65. For any participant who was unable to sense above 6.65, we applied the score of 6.65 in the analysis. Lower scores indicate a better outcome.
Time Frame: as for outcome 1
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Cutaneous Sensory Touch Threshold using Semmes-Weinstein Monofilaments Score for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
Scores on a scale
  Baseline | 4.17 [3.42 to 5.62]
  Post-Intervention: number analyzed (Participants) | 2
  Post-Intervention | 3.72 [3.09 to 4.34]
  3m follow-up | 4.24 [3.35 to 5.88]

6. Secondary Outcome: Stroke Impact Scale (SIS)
Description: The SIS is a 59 item measure of strength, hand function, activities of daily living, mobility, communication, emotion, memory, and participation. Each item is rated in a 5 point scale in terms of difficulty experienced in completing the item, ranging from 1 (could not do it at all) to 5 (not difficult at all).
  We reported here the total of strength (minimum possible score 4 and maximum possible score 20) and hand portion (minimum possible score 5 and maximum possible score 25). Subscale scores were summed to compute the total score (minimum possible score 9 and maximum possible score 45). Decimals are included in the lower and upper limits of the Full Range in the "baseline" row as these resulted from the averaging of two baseline scores.
Time Frame: as for outcome 2
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Stroke Impact Scale (SIS) Data for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  baseline | 21.83 [15.5 to 27.5]
  post-intervention: number analyzed (Participants) | 2
  post-intervention | 25 [23 to 27]
  3 month follow-up | 21 [16 to 26]

7. Secondary Outcome: Action Research Arm Test (ARAT)
Description: The ARAT test is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). ARAT is a validated quick (within ten to fifteen minutes) assessment of the paretic arm's functional disabilities, which offers uncomplicated and comprehensive feedback on the function of their arm, hand and fingers. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points. Higher scores indicate better performance. Decimals are included in the lower and upper limits of the Full Range in the "baseline" row as these resulted from the averaging of two baseline scores.
Time Frame: as for outcome 1
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Action Research Arm Test (ARAT) Data for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  Baseline | 29.6 [22.3 to 37.5]
  Post-intervention: number analyzed (Participants) | 2
  Post-intervention | 50 [43 to 57]
  3m follow-up | 43 [31 to 57]

8. Secondary Outcome: Chedoke McMaster Stroke Assessment (CMSA) Hand Subscale
Description: This test evaluate the stage of motor recovery for the paretic hand. Scores range from 0-7, with 7 representing full function of the hand.
Time Frame: as for outcome 2
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Chedoke McMaster Stroke Assessment (CMSA) Hand Subscale Data for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  Baseline | 3.5 [3 to 4]
  post-intervention: number analyzed (Participants) | 2
  post-intervention | 4.5 [4 to 5]
  3 month follow-up | 4 [4 to 4]

9. Secondary Outcome: Revised Nottingham Sensory Assessment: Kinaesthesia Subscale
Description: The kinaesthesia subscale measures an individuals ability to sense movement, direction of movement, and position sense at a given joint. The assessment involves the tester initiating passive movement in the individuals affected finger, wrist, elbow, and shoulder; while the individual attempts to match those movement with their opposite extremity. Scores for each joint range from 0-3, with higher scores meaning a better outcome.
  0 - Absent - no appreciation of movement taking place
  1. - appreciation of movement taking place
  2. - direction of movement sense
  3. - joint position sense The minimum score is 0 and the maximum score is 12. Decimals are included in the lower and upper limits of the Full Range in the "baseline" row as these resulted from the averaging of two baseline scores.
Time Frame: as for outcome 2
Population: Three right hand dominant participants who have chronic stroke (>1y) with moderate impairment at left side. Revised Nottingham Sensory Assessment: Kinaesthesia Subscale Data for the post-intervention could not be collected for 1 participant (DEV43).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Home Based Group
Number analyzed (Participants) | 3
scores on a scale
  baseline | 7.17 [4 to 9.5]
  post-intervention: number analyzed (Participants) | 2
  post-intervention | 8.5 [5 to 12]
  3 month follow-up | 7.6 [5 to 10]

ADVERSE EVENTS:
Time Frame: Adverse event data for the entire study was collected over 1 year, 10 months. For participant DEV14, adverse event data was collected for up to 11 months due to restrictions placed on the lab due to the COVID-19 pandemic (participant was not brought in for a 3 month follow-up but instead a 6 month follow-up). For DEV43 and DEV201, adverse event data was collected for up to 7 months.
Arm/Group | Home Based Group
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Limitations of the study:

1. This is a small size clinical trial, only 3 participants were recruited.
2. Due to the COVID-19 pandemic, deviations from the protocol were necessary to ensure safety. For one subject, post-intervention data could not be collected and for another, the 3 month follow-up data could not be collected.
3. For one secondary outcome measure, technical problems with measurement were encountered leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT03986216/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT03986216/SAP_001.pdf
  • Informed Consent Form (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03986216/ICF_002.pdf